CLINICAL TRIAL: NCT04472208
Title: Evaluation Clinical Study Of The Ambulatory Monitoring Solution (AMS)
Brief Title: AMS Evaluation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 123.04-2017-GES-0005
Record Dates: First submitted 2020-07-08; First posted 2020-07-15 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Patient Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ambulatory Monitoring Solution (Experimental): The evaluable device is a secondary monitoring device and no decisions/diagnosis will be made from these devices.
  Interventions: Device: Ambulatory monitoring solution

INTERVENTIONS:
Device: Ambulatory monitoring solution — Subjects participating in this study will be monitored with the site's standard of care primary monitor and the evaluable device as the secondary monitor.

SUMMARY:
A study to evaluate the operational and functional features of the Ambulatory Monitor Solution (AMS) as well as the ease of use of the system.

DETAILED DESCRIPTION:
The study is going to be conducted to collect feedback from the users about operation of AMS collect parameter raw data from patients in hospital ward setting using the investigational system for use in current and future AMS engineering and regulatory purposes as deemed appropriate by the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 years or older (≥18 years);
2. Able and willing to provide written informed consent independently.

Exclusion Criteria:

1. Have previously participated in this study (no subject may participate more than once);
2. Have an implantable pacemaker;
3. Diagnosed with infection requiring isolation; OR
4. Known to be pregnant and/or breast feeding;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
User feedback survey about the use of the Ambulatory Monitoring Solution | 5 days
  The feedback from the clinical users about operational features, alarms, user experience and ease of use of Ambulatory Monitoring Solution will be collected.

OTHER OUTCOMES:
Collect number of adverse events (AEs), serious adverse events (SAEs), and device issues | 1 year
  The safety objective is to collect safety information, including type and number of adverse events (AE), serious adverse events (SAE), and device issues. The descriptive statistical methods will be used to analyze AE and SAE data.

CONTACTS AND LOCATIONS:
Overall Officials: Meera Joshi, MBBS, Principal Investigator — St. Marys Hospital, London
Locations (1):
- Chelsea and Westminster Hospital, London, United Kingdom